CLINICAL TRIAL: NCT06859437
Title: Prevention of Clostridium Difficile Infections Using Lactobacillus Plantarum 299v Strain in Nephrology and Transplantation Department
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SilesianMUKB1/78/24
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Clostridioides Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LP299v group (Experimental): Participants: one capsule of LP299v orally per a day during the entire period of antibiotic therapy.
  Interventions: Dietary Supplement: Prevention of C. difficile infections using LP299v strain LP299v
- Placebo group (Placebo Comparator): Participants: one capsule of placebo orally per a day during the entire period of antibiotic therapy.
  Interventions: Dietary Supplement: Prevention of C. difficile infections using LP299v strain Placebo

INTERVENTIONS:
Dietary Supplement: Prevention of C. difficile infections using LP299v strain Placebo — Patients treated with antibiotics and at high CDI risk (patients after organ transplantation or receiving immunosuppressive therapy for any other reason) will be enroll to study.
  One capsule of placebo orally per a day during the entire period of antibiotic therapy.
  Arms: Placebo group
Dietary Supplement: Prevention of C. difficile infections using LP299v strain LP299v — Patients treated with antibiotics and at high CDI risk (patients after organ transplantation or receiving immunosuppressive therapy for any other reason) will be enroll to study.
  One capsule of LP299v orally per a day during the entire period of antibiotic therapy.
  Arms: LP299v group

SUMMARY:
The aim of this study was to analyze whether the use of the LP299v strain reduces the risk of Clostridium difficile infection (CDI) among patients receiving antibiotics and hospitalized in the nephrology and transplantation ward.

Adutt patients from risk group (receiving immunosuppressive drugs and treated with antibiotics) were enrolled into study.

Patients who meet the above criteria for inclusion in the study will be assigned to one of two groups. Patients in group I (study) will receive a probiotic containing the Lactobacillus plantarum 299v strain of bacteria as part of the prophylaxis of Clostridioides difficile infection. The daily dose is 1 capsule containing approximately 10x109 colony-forming units of live bacteria taken orally with a meal. Patients in group II (control) will receive a placebo. The duration of probiotic or placebo use will be 3 months. Assignment to groups I and II will be random. The number of patients in each group will be 150.

Participants will be divided into two groups. First group will receive one capsule of Lactobacillus plantarum 299v (LP299v) orally per a day. Second group will receive placebo. The observation period will last 3 months. The evaluation will consist of an interview, physical examination and laboratory tests.

DETAILED DESCRIPTION:
The study is prospective. It will include 300 patients undergoing antibiotic therapy. The duration of the study is estimated at 36 months (from 01.10.2024 to 31.10.2027).

The study will be conducted among patients hospitalized in the Clinic of Nephrology, Transplantology and Internal Medicine of the Medical University of Silesia/Department of Nephrology, Transplantology and Internal Medicine of the Independent Public Clinical Hospital named after Andrzej Mielęcki of the Medical University of Silesia in Katowice. The study will include patients undergoing immunosuppressive treatment undergoing antibiotic therapy. The exclusion criterion from the study is the lack of consent of the patient to participate in the study.The aim of this study was to analyze whether the use of the LP299v strain reduces the risk of Clostridium difficile infection (CDI) among patients receiving antibiotics and hospitalized in the nephrology and transplantation ward.

Adutt patients from risk group (receiving immunosuppressive drugs and treated with antibiotics) were enrolled into study.

Patients who meet the above criteria for inclusion in the study will be assigned to one of two groups. Patients in group I (study) will receive a probiotic containing the Lactobacillus plantarum 299v strain of bacteria as part of the prophylaxis of Clostridioides difficile infection. The daily dose is 1 capsule containing approximately 10x109 colony-forming units of live bacteria taken orally with a meal. Patients in group II (control) will receive a placebo. The duration of probiotic or placebo use will be 3 months. Assignment to groups I and II will be random. The number of patients in each group will be 150.

Participants will be divided into two groups. First group will receive one capsule of Lactobacillus plantarum 299v (LP299v) orally per a day. Second group will receive placebo. The observation period will last 3 months. The evaluation will consist of an interview, physical examination and laboratory tests.

The patient interview will include, among others:

* assessment of gastrointestinal complaints
* assessment of the number of stools per day and their consistency
* incidence of CDI
* incidence of other infectious diseases

The following laboratory and microbiological tests are planned for all patients in the randomized study:

* microbiological assessment of stool before starting treatment
* measurement of C-reactive protein, interleukin 6 and lipopolysaccharide LPS concentration in blood serum and assessment of peripheral blood morphology before starting treatment, on the 7th day of treatment and after 1 month.
* blood culture on MRS Agar before starting treatment, on the 8th-10th day of treatment and after 1 month After 3 months, a telephone interview with the patient is planned to collect information about the occurrence of diarrhea or other gastrointestinal disorders, Clostridioides difficile infection or other infectious diseases in the period of 3 months from the start of probiotic or placebo use.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* organ transplantation or receiving immunosuppressive drugs for any other reasons
* antibiotics therapy

Exclusion Criteria:

* no consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Clostridium difficile infection | Three month

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Transplantation and Intenal Medicine Medical University of Silesia, Poland, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided